CLINICAL TRIAL: NCT00089180
Title: A Phase IIb Randomized, Double-Blind, Placebo-Controlled Clinical Trial of Topical Bacteriophage T4 Endonuclease V in Renal Allograft Recipients With a History of Non-melanoma Skin Cancer
Brief Title: T4N5 Liposomal Lotion in Preventing The Recurrence of Nonmelanoma Skin Cancer in Patients Who Have Undergone a Kidney Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2012-02619; UAB-0323; CDR0000378098; N01CN15136 (Other Grant/Funding Number: US NIH Grant/Contract Award Number)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2013-06

CONDITIONS: Actinic Keratosis; Basal Cell Carcinoma of the Skin; Recurrent Skin Cancer; Squamous Cell Carcinoma of the Skin
MeSH Terms: conditions — Keratosis, Actinic; Carcinoma, Basal Cell; Skin Neoplasms | interventions — Deoxyribonuclease (Pyrimidine Dimer); endonuclease V, phage T4

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (liposomal T4N5 lotion) (Experimental): Patients apply T4N5 liposomal lotion topically to non-occluded, sun-exposed areas of the head, neck, face, and upper extremities once daily for 12 months.
  Interventions: Drug: liposomal T4N5 lotion; Other: laboratory biomarker analysis
- Arm II (placebo) (Placebo Comparator): Patients apply placebo topically to non-occluded, sun-exposed areas of the head, neck, face, and upper extremities once daily for 12 months.
  Interventions: Other: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: liposomal T4N5 lotion — Given topically
  Other Names: bacteriophage T4 endonuclease V in liposomal lotion; Dimericine; T4 endonuclease V liposomal lotion; T4N5 liposomal lotion
  Arms: Arm I (liposomal T4N5 lotion)
Other: placebo — Given topically
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well T4N5 liposomal lotion works in preventing the recurrence of nonmelanoma skin cancer in patients who have undergone a kidney transplant. Chemoprevention therapy is the use of certain drugs to try to prevent the development of or recurrence of cancer. T4N5 liposomal lotion may be effective preventing the recurrence of nonmelanoma skin cancer in patients who have undergone a kidney transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the incidence of nonmelanoma skin cancer (NMSC) (average per patient) on the sun-exposed skin of renal transplant recipients with a history of NMSC treated with T4N5 liposomal lotion vs placebo.

SECONDARY OBJECTIVES:

I. Compare the proportion of these patients who develop NMSC on sun-exposed skin during treatment and after cessation of treatment with these regimens.

II. Compare the incidence of NMSC on the sun-exposed skin of these patients after cessation of treatment with these regimens.

III. Compare the incidence of recurrent and de novo actinic keratoses (AKs) in patients treated with these regimens.

IV. Determine whether either of these regimens induces regression of AKs left untreated on the sun-exposed skin of these patients.

V. Compare the proportion of these patients who develop melanoma, in both treated and untreated sites, during and after cessation of treatment with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to study center. Patients are randomized to 1 of 2 arms.

Six months before randomization, lesions suspicious for nonmelanoma skin cancer (NMSC) are surgically removed and histologically analyzed. All but 10 randomly selected non-suspicious lesions are removed. Of these 10 lesions, 5 are shave biopsied immediately pre-treatment for histologic and surrogate endpoint biomarker (SEB) analysis and to determine a baseline actinic keratosis: wart ratio. Patients also undergo a pre-treatment biopsy of normal appearing sun-exposed and non-sun-exposed skin (buttocks).

Arm I: Patients apply T4N5 liposomal lotion topically to non-occluded, sun-exposed areas of the head, neck, face, and upper extremities once daily for 12 months.

Arm II: Patients apply placebo topically to non-occluded, sun-exposed areas of the head, neck, face, and upper extremities once daily for 12 months.

Treatment in both arms continues in the absence of the development of metastatic cutaneous squamous cell cancer or melanoma. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study within 6 months.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically confirmed nonmelanoma skin cancer
* Renal transplant recipient ≥ 4 years ago

  * Currently receiving standard multi-agent pharmacologic immunosuppression
* Fitzpatrick skin type I, II, or III
* Sun-damaged skin with ≥ 10 lesions consistent with actinic keratoses OR wart on the upper extremities (arms, forearms, hands), neck, face, and exposed scalp combined
* No history of keloid formation
* No known photosensitivity disorder
* No history of malignant melanoma
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No diagnosis of acute allograft rejection within the past 30 days requiring an increase in immunosuppression
* No invasive malignancy within the past 4 years except curatively excised NMSC, cured polyclonal posttransplantation lymphoproliferative disease, carcinoma in situ of the cervix, stage 0 chronic lymphocytic leukemia, unless all of the following criteria are met:

  * No current evidence of disease
  * No treatment for the invasive malignancy within the past 6 months
  * No concurrent or planned therapy for the invasive malignancy
  * Has an expected disease-free survival of at least 5 years
* No diagnosis of melanoma or melanoma in situ
* No other medical or psychosocial condition that would preclude study participation
* No likelihood, in the opinion of the transplant surgeon/nephrologist, to experience graft loss and/or discontinue standard immunosuppressive therapy during study treatment
* More than 30 days since prior and no concurrent topical chemotherapy (including topical fluorouracil) to areas being studied
* No concurrent topical preparations containing corticosteroids
* More than 30 days since prior and no concurrent local radiotherapy to a study area
* More than 30 days since prior and no concurrent cryotherapy to target lesions
* No prior or concurrent experimental immunosuppressive agents
* More than 30 days since prior investigational medication
* More than 30 days since prior and no concurrent systemic psoralens or retinoids
* More than 60 days since prior and no concurrent laser resurfacing, dermabrasion, or chemical peels to a study area
* No other concurrent investigational agents
* No other concurrent topical medications, including prescription and over the counter preparations, to the areas being studied (e.g., upper arms, forearms, neck, face, and scalp)

  * Concurrent moisturizer, emollient, and sunscreen allowed
* No concurrent topical preparations containing vitamin A derivatives
* No concurrent nonsteroidal anti-inflammatory drugs

  * Concurrent cardioprotective doses of aspirin (< 100 mg/day) allowed

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-03; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Incidence of nonmelanoma skin cancer (NMSC) | Up to 18 months
  Descriptive statistics such as mean, median, standard deviation will be calculated to summarize the number of new NMSC for each of the two randomization arms and compared using the Wilcoxon rank-sum test.

SECONDARY OUTCOMES:
Proportion of patients who develop NMSC during and after completion of study therapy | Up to 18 months
  Calculated for the study drug and placebo arms and compared using the Fisher's exact or chi-square test.
Incidence of NMSC | Up to 18 months
  Summarized by treatment arm and compared using the Wilcoxon rank-sum test.
Incidence of recurrent and de novo actinic keratoses (AKs) after completion of study therapy | Up to 18 months
  Summarized by treatment arm and compared using the Wilcoxon rank-sum test. Similarly, multivariate Poisson regression model will be utilized to compare the cumulative number of incident AKs at the end of treatment as a function of treatment arm and covariates.
Number of regressed AKs after completion of study therapy | At 18 months
  Summarized by treatment group and compared using the Wilcoxon rank-sum test. Similarly, multivariate Poisson regression model will be utilized to compare the cumulative number of regressed AKs at the end of treatment as a function of treatment group and covariates. In addition to the covariates listed above, the number of AKs at baseline will be included as a covariate in the model.
Risk of developing melanoma in both treated and untreated sites | Up to 18 months
  The data will be collected and analyzed by scoring both total body melanoma distribution and those in lotion treatment sites. Relative risk will be calculated for the development of melanomas. The Chi-Square test will be used to explore the risk relationships.
Change in SEBs levels | From baseline to 12 months
  Descriptive statistics will be calculated at baseline and end of treatment for several SEBs by treatment arm. The change in SEB levels will be also calculated for each patient and compared between treatment arms using either the two-sample t-test or Wilcoxon rank-sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Elmets, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Comprehensive Cancer Center, Birmingham, Alabama, United States